CLINICAL TRIAL: NCT06681454
Title: Retrospective Comparative Cohort Analysis of Darn and Lichtenstein Repair Methods for Bilateral Inguinal Hernias in Adult Males in a Low-Resource Setting: a Single-Centre Study in Sudan
Brief Title: Comparing Darn and Lichtenstein Repair for Bilateral Inguinal Hernias in Adult Males in a Low-Resource Setting
Status: Completed | Type: Observational
Sponsor: Sudan Medical Specialization Board (Other Government)
Collaborators: Sudan Medical Specialization Board (SMSB) (Other Government)
Responsible Party: Principal Investigator, Alsadig Suliman, General surgery, Federal Ministry of Health, Sudan
Other Study IDs: SMSB-HERNIA-001-2024; SMSB-HERNIA-001-2024 (Registry Identifier: Inguinal Hernia Repair Methods Study Registry)
Record Dates: First submitted 2024-10-24; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Darn Vs. Lichtenstein Hernia Outcomes; Outcomes of Darn and Lichtenstein Hernia Repairs; Bilateral Inguinal Hernia: Darn Vs. Lichtenstein
Keywords: Retrospective cohort study; Low-resource setting; Medical records analysis; Bilateral inguinal hernia; Lichtenstein repair method; Darn repair method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lichtenstein Repair Cohort: This group consists of adult male patients who underwent bilateral inguinal hernia repair using the Lichtenstein technique. The Lichtenstein method involves the use of a synthetic mesh to provide support to the weakened abdominal wall, minimizing the risk of recurrence and promoting quicker recovery.
- Darn Repair Cohort: This group comprises adult male patients who underwent bilateral inguinal hernia repair using the Darn technique. The Darn method is a tension-free repair technique that utilizes the patient's own tissue without the use of mesh, aimed at reducing postoperative pain and complication rates.

SUMMARY:
This retrospective study evaluates the efficacy of Darn versus Lichtenstein repair methods in treating bilateral inguinal hernias in adult males within a low-resource setting in Sudan. The study aims to determine which surgical technique results in better postoperative outcomes, focusing on complication rates, recurrence, and recovery times. Data for this analysis will be sourced from medical records of patients who underwent these procedures between January 2021 and October 2023 at Al-Waleedeen Specialized Hospital.

DETAILED DESCRIPTION:
Study Design and Setting

This is a retrospective comparative cohort study undertaken at Al-Waleedeen Specialized Hospital, a governmental tertiary care center in Gezira State, Sudan. The study period spans from January 2021 to October 2023, involving adult males diagnosed with bilateral inguinal hernias.

Study Procedures

Medical records will be systematically reviewed to extract data on surgical technique employed-either Darn or Lichtenstein method. The review will document specific procedural details such as the type of anesthesia used, duration of the surgeries, surgical team composition, and intraoperative management techniques. Information on immediate postoperative care will also be collected, focusing on pain management strategies and mobilization protocols.

Data Collection

The data collection will emphasize capturing precise measures related to surgical outcomes. This includes the exact nature and timing of any postoperative complications (e.g., infection, hematoma, seroma), the precise time to recurrence if applicable, and detailed recovery timelines including return to daily activities and work. All data points will be aligned with the definitions set forth in the STROBE guidelines to maintain consistency and reliability in reporting.

Analytical Methods

The primary analytical approach will involve comparing the frequency and severity of complications between the two surgical methods. Statistical methods will include chi-square tests for categorical data and t-tests for continuous variables, with a significance level set at p<0.05. Kaplan-Meier curves may be used to estimate recurrence rates over the follow-up period, and a Cox proportional hazards model will assess risk factors for recurrence and complications.

Outcome Measures

The main outcome measures will focus on:

Short-term complications within the first three months post-surgery. Long-term hernia recurrence over the follow-up period. Recovery timelines, quantified by time until return to usual activities and work.

Ethical Considerations

The study protocol has been reviewed and approved by the Institutional Review Board at Al-Waleedeen Specialized Hospital. All data will be de-identified to ensure confidentiality and compliance with ethical standards for research involving human subjects.

ELIGIBILITY:
Inclusion Criteria:

Male patients aged 16 to 85 years. Diagnosed with bilateral primary direct or indirect inguinal hernias. Underwent open elective repairs using either the Lichtenstein or Darn method.

Exclusion Criteria:

Patients with recurrent hernias. Female patients. Patients with unilateral hernias. Those undergoing laparoscopic or emergency surgery. Patients with poorly controlled diabetes (A1C > 7). Patients diagnosed with cancer, tuberculosis. Patients with giant inguinoscrotal hernias.

Ages: 16 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This indicates that eligibility is limited by biological sex, as the study is focused on adult male patients for the surgical techniques being analyzed
Study Population: The study population will consist of adult male patients aged 16 to 85 years who present with bilateral primary direct or indirect inguinal hernias at Al-Waleedeen Specialized Hospital in Gezira State, Sudan. Participants will be selected based on their medical records and will have undergone open elective hernia repair using either the Darn or Lichtenstein technique during the recruitment period from January 2021 to October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Complication Rates | Up to 3 months post-surgery
  Number of patients experiencing postoperative complications. Unit of Measure: Percentage of total patients.
Hernia Recurrence Rates | Up to 3 months post-surgery .
  Number of patients with recurrence of hernia after initial repair. Unit of Measure: Percentage of total patients.

SECONDARY OUTCOMES:
Postoperative Pain Level | Assessed at 24 hours, 72 hours, and 1 week post-surgery.
  Average pain scores reported by patients using the Visual Analog Scale. Unit of Measure: Pain score on a scale from 0 (no pain) to 10 (worst possible pain).
Duration of Hospital Stay | From date of surgery to discharge, within 30 days post-surgery
  Length of hospital stay post-surgery. Unit of Measure: Number of days from surgery to discharge.
Recovery Times | Assessed at 2 weeks, 1 month, and 3 months post-surgery.
  Time taken for patients to return to usual activities/work post-surgery. Unit of Measure: Number of days from surgery to return to usual activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Waleedeen Specialized Hospital, Wad ALnaeem, Gazira, Sudan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to several considerations. First, the data includes sensitive personal health information, which must be protected to comply with privacy regulations and ethical standards. Additionally, the study is conducted in a low-resource setting, where data management and sharing capabilities may be limited. Ensuring the confidentiality and anonymity of participants is paramount, and sharing IPD could compromise these ethical obligations. Finally, the data will be used exclusively for the purpose of this study to inform clinical practice within the context of the local healthcare system, rather than for broader dissemination.